CLINICAL TRIAL: NCT06618703
Title: Endocrine Follow-up After Cerebral Radiotherapy Performed Before Age 16 (Direct Cerebral Field or Following Facial, Cervical or High Ear, Nose, and Throat Radiotherapy)
Brief Title: Brain Irradiation for Childhood Cancer - Endocrine Monitoring During the First Years
Acronym: BIChE-1
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Angers (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 49RC24_0193
Record Dates: First submitted 2024-07-30; First posted 2024-10-01 (Actual); Last update posted 2025-02-25 (Actual); Status verified 2025-02

CONDITIONS: Endocrine; Deficiency; Hypothalamo-Pituitary Disorder; Radiotherapy Side Effect
Keywords: Hypothalamic-pituitary axis deficiency; cerebral radiotherapy; brain tumours; endocrine monitoring; follow-up protocol
MeSH Terms: conditions — Radiation Injuries; Brain Neoplasms | interventions — Blood Specimen Collection

STUDY DESIGN:
Intervention Model Description: Intervention research with minimum risks and constraints
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Study Arm (Experimental): Specific interventions:
  For all patients, an insulin level is added every 2 years. For patients under 8 years of age, additional elements such as testosterone (in male patients), Luteinizing hormone , Follicle-stimulating hormone, estradiol (in female patients), inhibin B +/- Anti-Müllerian hormone are measured during the usual blood test.
  A urinary check-up is systematically added for all patients, whereas it is usually only prescribed after certain chemotherapies (platinum salts, ifosfamide), nephrectomy, radiotherapy to the flanks as part of routine care. This check-up will be carried out at 2 and 4 years post-radiotherapy.
  For patients aged 12 and over, a second bone densitometry is performed at the end of follow-up, even if the first is normal. In routine care, international guidelines recommend this first bone densitometry, and the second is usually performed only if the first was abnormal.
  Interventions: Radiation: Blood sample, urine sample, osteodensitometry

INTERVENTIONS:
Radiation: Blood sample, urine sample, osteodensitometry — Blood sample, urine sample, osteodensitometry

SUMMARY:
BICHE- 1: Brain Irradiation for Childhood cancer - Endocrine monitoring during the first five years is a study of endocrine monitoring after cerebral radiotherapy.

The study concerns patients in remission at the end of oncological treatment aged between 4 and 18 years at the time of inclusion and who have had radiotherapy before the age of 16, irradiating all or part of the brain, with a delay between the end of radiotherapy and inclusion of less than 5 years. Patients will be included during a routine visit to the paediatric endocrinologist.

The protocol for the Biche 1 study has been designed and discussed in a multidisciplinary and multicentre manner, based on data from the literature and the French reference document (September 2021) "National protocol for diagnosis and care - congenital pituitary deficiency".

In this population, the investigators will conduct a descriptive and exploratory study to establish recommendations for medium-term follow-up; to improve screening for endocrine deficiencies affecting the hypothalamic-pituitary axis in order to improve patients' quality of life and state of health; and to better define dose-volume constraints on the axis.

The study will also focus on better detection and characterisation of chronic fatigue as a potential sequela of pituitary deficiencies, in particular by means of a questionnaire assessing fatigue (PedsQL Multidimensional Fatigue scale) which will also be systematically administered and completed annually.The expected sample size is 100-150 patients treated for a brain tumour and 60-80 patients treated for another tumour but with an irradiation field covering all or part of the brain.

ELIGIBILITY:
Inclusion Criteria:

* Patient aged 4 years or more (≥4) and less than 18 years (<18) at inclusion
* Treated with radiotherapy to part or all of the brain for cancer or hematological malignancy before age 16 (≤15)
* Post-radiotherapy time less than or equal to 5 years (≤5)
* In remission of this pathology at the end of oncological treatments, or, with stable residual disease without treatment for 2 years or more (≥2)
* Signature of informed consent from parents or legal guardian
* Patient affiliated to the social security system or beneficiary of such a system

Exclusion Criteria:

* Patients who have relapsed or developed a second cancer with a post-treatment delay of < 1 year
* Patient in palliative situation
* Brain irradiation with dosimetric data showing sparing of the hypothalamic-pituitary axis (Dmax hypothalamic-pituitary axis < 15 Gy)
* Patient with a known hypothalamic-pituitary axis endocrine deficit prior to radiotherapy
* Refusal of child or parents

Ages: 4 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 230 (Estimated)
Dates: Start 2025-03 (Estimated); Primary Completion 2030-10 (Estimated); Study Completion 2030-10 (Estimated)

PRIMARY OUTCOMES:
Endocrine toxicities assessment after radiotherapy involving all or part of the brain in children, adolescents and young adults treated for cancer before the age of 16 (≤15 years) | Follow-up of 4 years, within a maximum of 5 years post-radiotherapy
  Measurement of hormon level for :
  * growth hormone deficiency
  * gonadal insufficiency
  * hypothyroidism
  * adrenal insufficiency

SECONDARY OUTCOMES:
To define risk factors for anterior pituitary insufficiency in patients who received brain radiotherapy, taking into account treatment characteristics and clinical data. | Follow-up of 4 years, within a maximum of 5 years post-radiotherapy
  Dose absorbed (Gy) by sensitive organs: This parameter corresponds to the total amount of radiation absorbed by the hypothalamus and pituitary gland, two key structures of the endocrine axis. A cumulative dose above certain thresholds is associated with a higher risk of long-term endocrine dysfunction - possibly after adjustment for the biological equivalent dose (which also takes fractionation into account).
To define risk factors for anterior pituitary insufficiency in patients who received brain radiotherapy, taking into account treatment characteristics and clinical data. | Follow-up of 4 years, within a maximum of 5 years post-radiotherapy
  Maximum dose (Dmax): The maximum dose received by a small portion of tissue in these critical organs.
To define risk factors for anterior pituitary insufficiency in patients who received brain radiotherapy, taking into account treatment characteristics and clinical data. | Follow-up of 4 years, within a maximum of 5 years post-radiotherapy
  Volume irradiated (%): This parameter measures the proportion of the organ exposed to radiotherapy.
To define risk factors for anterior pituitary insufficiency in patients who received brain radiotherapy, taking into account treatment characteristics and clinical data. | Follow-up of 4 years, within a maximum of 5 years post-radiotherapy
  Average dose (Dmean) and D50%: The average and median dose received by the whole organ.
To define risk factors for anterior pituitary insufficiency in patients who received brain radiotherapy, taking into account treatment characteristics and clinical data. | Follow-up of 4 years, within a maximum of 5 years post-radiotherapy
  Minimum dose (Dmin): minimum dose received by the organ.
To define risk factors for anterior pituitary insufficiency in patients who received brain radiotherapy, taking into account treatment characteristics and clinical data. | Follow-up of 4 years, within a maximum of 5 years post-radiotherapy
  Dose-volume histogram (DVH): The DVH analysis enables you to visualize the dose distribution over the entire organ, and to identify any thresholds other than those listed above.
Hormone deficiencies on fatigue in adult patients | Follow-up of 4 years, within a maximum of 5 years post-radiotherapy
  Measurement by a questionnaire assessing fatigue (PedsQL Multidimensional Fatigue scale) composed of 18 items comprising 3 dimensions.
  5-point Likert scale from: 0 (Never) to 4 (Almost always) 3-point Likert scale from: 0 (Not at all), 2 (Sometimes) and 4 (A lot) for the Child Report for Young Children (ages 5-7) then Items are reverse scored and linearly transformed to a 0-100 scale as follows: 0=100, 1=75, 2=50, 3=25, 4=0
Hormone deficiencies on cognitive disorders in adult patients | Follow-up of 4 years, within a maximum of 5 years post-radiotherapy
  Measurement by a questionnaire assessing fatigue (PedsQL Multidimensional Fatigue scale) composed of 18 items comprising 3 dimensions.
  5-point Likert scale from: 0 (Never) to 4 (Almost always) 3-point Likert scale from: 0 (Not at all), 2 (Sometimes) and 4 (A lot) for the Child Report for Young Children (ages 5-7) then Items are reverse scored and linearly transformed to a 0-100 scale as follows: 0=100, 1=75, 2=50, 3=25, 4=0
Fatigue measurement in patients after the introduction of hormone replacement therapy | Follow-up of 4 years, within a maximum of 5 years post-radiotherapy
  Measurement by a questionnaire assessing fatigue (PedsQL Multidimensional Fatigue scale) composed of 18 items comprising 3 dimensions.
  5-point Likert scale from: 0 (Never) to 4 (Almost always) 3-point Likert scale from: 0 (Not at all), 2 (Sometimes) and 4 (A lot) for the Child Report for Young Children (ages 5-7) then Items are reverse scored and linearly transformed to a 0-100 scale as follows: 0=100, 1=75, 2=50, 3=25, 4=0